CLINICAL TRIAL: NCT04316351
Title: Efficacy and Safety of Toripalimab (JS001) Combined With Pemetrexed and Anlotinib for Patients With T790M Positive Non-Small Cell Lung Cancer After Osimertinib Resistance：a Phase II,Muti-center, Single Arm Study
Brief Title: Efficacy and Safety of Toripalimab (JS001) Combined With Pemetrexed and Anlotinib for Patients With T790M Positive Non-Small Cell Lung Cancer After Osimertinib Resistance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Chief Physician, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC2002
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: IIIb/IV NSCLC With T790M Positive Mutations Failed to Osimertinib Therapy
MeSH Terms: interventions — toripalimab; Pemetrexed; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab + Pemetrexed + Anlotinib (Experimental)
  Interventions: Drug: Toripalimab + Pemetrexed + Anlotinib

INTERVENTIONS:
Drug: Toripalimab + Pemetrexed + Anlotinib — Toripalimab 240 mg iv d1 + anlotinib 12mg po d1-d14 + pemetrexed 500mg / m2 d1 Q3W for 4 cycles, followed by Toripalimab 240mg iv d1 + anlotinib 12mg po d1 + pemetrexed 500mg / m2 d1 Q3W for another 31 cycles (up to a total of 35 cycles).
  If there is no disease progression, patients will receive anlotinib po 12mg d1-d14 + pemetrexed 500mg / m2 d1, Q3W for maintenance therapy until PD per RECIST v1.1 or loss of clinical benefit.
  Other Names: JS001

SUMMARY:
This is an open-label, single-arm, multi-center, phase II exploratory study that evaluates the efficacy and safety of Toripalimab injection (JS001) combined with Pemetrexed and Anlotinib as a second-line treatment for patients with T790M positive Non-Small Cell Lung Cancer (IIIb / IV ) after Osimertinib resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand this study and voluntarily sign the informed consent form (ICF);
2. Histologically and/or cytologically confirmed Stage IIIb / IV NSCLC (according to the seventh edition of AJCC); patients with T790M-positive mutations who were resistant to Osimertinib treatment;
3. At least one measurable lesion (according to RECIST 1.1); Note: Lesions that have previously received radiotherapy cannot be regarded as target lesions, unless the lesions clearly progress after radiotherapy;
4. Agree to provide formalin-fixed tumor specimens or biopsy specimens after the subject is diagnosed with metastatic cancer, at least 15 sections; if the recent biopsy is not feasible, allow to receive biopsy specimens before adjuvant/neo-adjuvant chemotherapy (archived specimens);
5. ECOG PS 0-2
6. Life expectancy ≥3 months.
7. The laboratory examination results within 7 days before enrollment must meet the following standards:

   1. Neutrophils ≥1.5 × 109 / L;
   2. Platelets ≥100 × 109 / L;
   3. Hemoglobin ≥90g / L (no infusion of concentrated red blood cells within 4 weeks);
   4. Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL / min;
   5. Total serum bilirubin ≤ 1.5 × ULN;
   6. AST and ALT ≤ 2.5 × ULN; in patients with liver metastases, ALT and AST ≤ 5 × ULN;
   7. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN unless the subject is receiving anticoagulant therapy; Activated partial thrombin time (aPTT) or partial thrombin time (PTT) ≤ 1.5 × ULN unless the subject is receiving anticoagulant therapy.
8. Women of childbearing age must confirm that the serum pregnancy test is negative and agree to use effective contraception during drug use and within 60 days after the last dose. Women of childbearing age are defined as sexually mature women in this program: 1) not undergoing hysterectomy or bilateral ovariectomy, 2) natural menopause has not continued for 12 months (amenorrhea after cancer treatment does not exclude fertility).

Exclusion Criteria:

1. Incorporate other driver gene mutations with known drug treatments, including but not limited to: ALK gene rearrangement, ROS1 mutation, BRAF600E mutation, etc .;
2. Received systemic chemotherapy for advanced NSCLC within 4 weeks before enrollment;
3. Have received EGFR-TKI treatment within 2 weeks before enrollment;
4. Received radiotherapy within 4 weeks or radiopharmaceutical treatment within 8 weeks before enrollment, except for local palliative radiotherapy for bone metastases;
5. Uncontrollable or symptomatic hypercalcemia (> 1.5mmol / L ionized calcium or calcium> 12 mg / dL or corrected serum calcium> ULN);
6. Have undergone major surgery or have not completely recovered from the previous operation within 4 weeks before enrollment ;
7. The toxicity of previous antitumor treatment has not recovered to CTCAE 0-1, except for hair loss；
8. Active or untreated CNS metastases detected by CT or MRI before screening and imaging evaluation: If a new asymptomatic CNS metastases is detected during the screening period , it must undergo radiation therapy and / or surgery . After treatment, if met all other criteria, no additional brain scan is required . Patients who have previously received brain or meningeal metastasis treatment and maintained clinical stability for at least 2 weeks, stopped systemic hormonal therapy (> 10 mg / day of prednisone or other equivalent hormones) for more than 2 weeks can be included;
9. Spinal cord compression that has not undergone radical surgery and / or radiation therapy, or previously diagnosed spinal cord compression with no clinical evidence showing that the disease is stable for ≥ 4 weeks before enrollment
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently);
11. have a history of idiopathic pulmonary fibrosis, organizing pneumonia (such as occlusive bronchiolitis), drug-induced pneumonia, idiopathic pneumonia, or have evidence of active pneumonia detected by chest CT;
12. Clinically uncontrolled active infections, including but not limited to acute pneumonia;
13. Past or present with other malignancies (except for non-melanoma skin basal cell carcinoma, breast / cervical carcinoma in situ, and other malignancies that have not been treated in the past five years and have been effectively controlled);
14. The patients have any active autoimmune disease or a history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism, reduced thyroid function; Patients with vitiligo or childhood asthma that have completely recovered and do not require any intervention in adults can be included; asthma with bronchodilators required for medical intervention cannot be included);
15. Known clinically significant liver diseases, including active viral hepatitis, alcoholic hepatitis or other hepatitis, cirrhosis, fatty liver, hereditary liver disease, uncontrollable major seizures, or superior vena cava syndrome;
16. Previously used anti-PD-1 antibody, anti-PD-L1 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell co-stimulation or checkpoint pathway).
17. Patients with active tuberculosis (TB) are receiving antituberculosis treatment or have received antituberculosis treatment within 1 year before screening;
18. After obtaining the approval of the clinical monitor, patients within 4 weeks before the first medication patients receiving systemic immunosuppressive drugs (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and TNF-α ) or receiving short-term, low-dose systemic immunosuppressive drugs or receiving one-time shock therapy with systemic immunosuppressive drugs (eg, 48 hours of glucocorticoid treatment for contrast allergic reactions) can be enrolled in the study. Patients receiving mineralocorticoids (such as fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible to participate in the study;
19. Have received any anti-infective vaccine (such as influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment;
20. A pregnant or lactating woman or a woman who may be pregnant have a positive pregnancy test before the first use of the drug; a patient with fertility who is unwilling to receive contraceptives or her sexual partner is unwilling to receive contraceptives;
21. History of HIV infection
22. Patients who had obvious hemoptysis (>50ml/day) within 3 months before enrollment; Patients who experienced bleeding symptoms of clinical significance or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc within 3 months before enrollment ;
23. Any other disease or condition of clinical significance that the investigator believes may affect protocol compliance, or affect the signing of an ICF, or is not suitable for participation in this clinical trial;
24. A history of severe allergies, allergies or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins;
25. Patients who are allergic to known biological drugs produced by Chinese hamster ovary cells, or citric acid monohydrate, sodium citrate dihydrate, mannitol, polysorbate (a component of the test drug);
26. Patients who have previously received an allogeneic stem cell or parenchymal organ transplant.
27. CT or MRI shows that tumor locate within a distance of less than 5 mm from the large vessels, or there is a central tumor that invades the local large blood vessels; or there are obvious pulmonary cavity or necrotic tumors;
28. Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate （ORR） | two years
  Defined as percentage of participants achieving complete response (CR) and partial response (PR) assessed by the Independent Review Committee (IRC) according to the RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | two years
  assessed by IRC and researchers based on RECIST 1.1
Overall survival (OS) | two years
  assessed by IRC and researchers based on RECIST 1.1
Disease Control Rate (DCR) | two years
  assessed by IRC and researchers based on RECIST 1.1
Duration of disease response (DOR) | two years
  assessed by IRC and researchers based on RECIST 1.1
overall incidence of adverse events (AE) | two years
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No